CLINICAL TRIAL: NCT04073498
Title: An Adaptive Design, Phase I/IIa, Open Label, Multicentre, Single Dose Escalation and Multiple Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Intravenous and Subcutaneous Doses of SerpinPC in Healthy Male Volunteers and Male Participants with Severe Haemophilia a or B with or Without Inhibitors
Brief Title: The Safety and Tolerability of SerpinPC in Healthy Men and in Men with Severe Blood Disorders (haemophilia a and B)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ApcinteX Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: AP-0101
Record Dates: First submitted 2019-08-13; First posted 2019-08-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia a; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 7 parts (Part 1a, Part 1b, Part 2, Part 3, Part 4, Part 5 and Part 6).
  Part 1a will be a single ascending dose study in 15 healthy male subjects. Part 1b will be a single ascending dose study in a minimum of 12 male patients with severe hemophilia A or B with or without inhibitors.
  Part 2 will involve subcutaneous doses not exceeding 1.2 mg/kg SerpinPC every 4 weeks in patients with severe hemophilia A or B with or without inhibitors.
  Part 3 will involve subcutaneous doses of SerpinPC in patients who have completed Week 24 of Part 2.
  Part 4 will involve subcutaneous doses of 1.2 mg/kg SerpinPC every 2 weeks for 24 weeks in patients who have completed Week 48 of Part 3.
  Part 5 will involve subcutaneous doses of 1.2 mg/kg SerpinPC every 2 weeks for 52 weeks for patients who have completed Week 24 of Part 4.
  Part 6 will involve a subcutaneous flat dose of 60mg SerpinPC every 2 weeks for 52 weeks for patients who have completed Week 52 of Part 5.
Who Masked: Participant
Masking Description: Part 1a: Open label for intravenous (IV) doses and single blinded for SC doses (subjects are blinded) Part 1b: Single blinded (patients are blinded) Part 2: Open label Part 3: Open label Part 4: Open label Part 5: Open label Part 6: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Part 1a - Cohort 1 (Experimental): A single IV infusion of 0.0003 mg/kg SerpinPC in healthy subjects.
  Interventions: Drug: SerpinPC
- Part 1a - Cohort 2 (Experimental): A single IV infusion of 0.001 mg/kg SerpinPC in healthy subjects.
  Interventions: Drug: SerpinPC
- Part 1a - Cohort 3 (Experimental): A single IV infusion of 0.003 mg/kg SerpinPC in healthy subjects.
  Interventions: Drug: SerpinPC
- Part 1a - Cohort 4 (Experimental): A single IV infusion of 0.01 mg/kg SerpinPC in healthy subjects.
  Interventions: Drug: SerpinPC
- Part 1a - Cohort 5 (Experimental): A single SC dose of 0.03 mg/kg SerpinPC and a single SC dose of placebo in healthy subjects.
  Interventions: Drug: SerpinPC; Drug: Placebo
- Part 1b - Cohort 6 (Experimental): A single SC dose of 0.1 mg/kg SerpinPC and a single SC dose of placebo in patients.
  Interventions: Drug: SerpinPC; Drug: Placebo
- Part 1b - Cohort 7 (Experimental): A single SC dose of 0.3 mg/kg SerpinPC and a single SC dose of placebo in patients.
  Interventions: Drug: SerpinPC; Drug: Placebo
- Part 1b - Cohort 8 (Experimental): A single SC dose of 0.6 mg/kg SerpinPC and a single SC dose of placebo in patients.
  Interventions: Drug: SerpinPC; Drug: Placebo
- Part 1b - Cohort 9 (Experimental): Two single SC doses of 0.6 mg/kg SerpinPC in patients.
  Interventions: Drug: SerpinPC
- Part 2 (Experimental): Up to 3 SC doses may be selected for Part 2 and each patient will be assigned a single SerpinPC dose level (and placebo). The dose for Part 2 will be determined from ongoing review of the Part 1 data. The dose in Part will not exceed 1.2 mg/kg, or the highest dose deemed safe from Part 1b.
  Interventions: Drug: SerpinPC; Drug: Placebo
- Part 3 (Experimental): A single flat SC dose of SerpinPC will be administered every 4 weeks for 48 weeks for patients who have completed Week 24 of Part 2. The dose level will be chosen after reviewing Part 2 data and will not exceed maximum dose level in Part 2.
  Interventions: Drug: SerpinPC
- Part 4 (Experimental): SC doses of 1.2 mg/kg SerpinPC will be administered every 2 weeks for 24 weeks for patients who have completed Week 48 of Part 3.
  Interventions: Drug: SerpinPC
- Part 5 (Experimental): SC doses of 1.2 mg/kg SerpinPC will be administered every 2 weeks for 52 weeks for patients who have completed Week 24 of Part 4.
  Interventions: Drug: SerpinPC
- Part 6 (Experimental): A single flat SC dose of 60mg SerpinPC will be administered every 2 weeks for 52 weeks for patients who have completed Week 52 of Part 5.
  Interventions: Drug: SerpinPC

INTERVENTIONS:
Drug: SerpinPC — Administered as IV infusion (over 30 minutes) or SC injection (abdomen) according to cohort dosing instructions.
Drug: Placebo — Matching placebo administered by SC injection according to cohort dosing instructions.
  Arms: Part 1a - Cohort 5; Part 1b - Cohort 6; Part 1b - Cohort 7; Part 1b - Cohort 8; Part 2

SUMMARY:
The purpose of this study is to investigate the safety and activity in the body of a new drug called SerpinPC.

The study will be split into 7 parts: Part 1a will be conducted in healthy male volunteers in the UK (up to 15) and Parts 1b, 2, 3, 4, 5 and 6 will be conducted in haemophilia A & B patients in Moldova and Georgia.

Part 1a of the study will look at how safe the drug is when given as single doses to healthy volunteers at different strengths and via 2 different routes of administration (through a vein or via an injection under the skin). Parts 1b, 2, 3, 4, 5 and 6 of the study will look at the safety of the drug when given as an injection under the skin to patients with severe haemophilia A or B.

The study will also investigate how the levels of the drug in the blood change over a period of time and how the drug acts in the body by taking blood samples. These blood samples will measure the concentration of the drug in the blood and measure certain aspects of the blood to determine how the drug affects them.

The study sponsor (ApcinteX) is developing this drug for the treatment of haemophilia A and haemophilia B, which are 2 types of rare blood disorders which affect the body's ability to form blood clots. Patients who have haemophilia A and B do not have certain clotting factors in their blood which means that they experience difficulty in stopping bleeding after injury and can be prone to extended periods of bleeding.

Current treatments for haemophilia involves injections which replace the missing factors in the blood. However these treatments are short term and therefore patients require regular treatments in order to manage the condition.

Therefore, there is a need to develop more effective treatments which provide longer term benefits. The aim of SerpinPC is to prevent bleeding rather than to have to treat bleeds to minimise pain and damage after they have occurred.

ELIGIBILITY:
Inclusion Criteria:

Part 1a (Healthy Subjects)

1. Males age ≥18 years and ≤55 years.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or delegate.
3. Willingness to give written consent to have data entered into The Over-volunteering Prevention System (TOPS).
4. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire trial.
5. Screening D-dimer ≤ 750 µg/L
6. Non-user of nicotine products i.e. non-smokers or ex-smokers who have stopped smoking or who had stopped using cigarette replacements for at least 6 months before the first dose of IMP.
7. Male subject willing to use 2 highly effective methods of contraception from the first dose administration until 3 months after dosing.
8. Subject with a body mass index (BMI) of 18 - 30 kg/m2 and weight ≥ 60 kg.
9. Subject with no clinically significant history of previous drug allergies.
10. Subject with no clinically significant abnormal Cytokine levels (IL6 and TNFα), serum biochemistry, haematology, coagulation and urinalysis within 28 days before the first dose of IMP.
11. Subject with negative urinary drugs of abuse (DOA) and alcohol screens, determined within 28 days before the first dose of IMP (N.B. A positive test result may be repeated at the Investigator's discretion).
12. Subject with negative human immunodeficiency virus (HIV), and hepatitis B surface antigen (HBsAg) and/or hepatitis C virus antibody (HCV Ab) test results at Screening.
13. Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before the first dose of IMP.
14. Subject with no clinically significant abnormalities in vital signs (supine blood pressure/pulse rate, oral temperature) determined within 28 days before the first dose of IMP.
15. Subject must be available to complete the study (including all follow up visits).
16. Subject must satisfy an Investigator about his fitness to participate in the study.

Part 1b and Part 2 (Patients)

1. Male age ≥18 years and ≤60 years.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the Investigator or delegate.
3. Patients with severe haemophilia (defined as having factor VIII/IX ≤ 0.02 IU/mL [2%]) with or without inhibitors, with an ABR (annualised bleeding rate) of 6 or more during the Observational Phase.
4. Patients on demand therapy with fVIII, fIX, rfVIIa (NovoSeven), FEIBA for treatment of bleeding.
5. Screening D-dimer ≤ 750 μg/L (DDU).
6. Adequate haematologic function, defined as having platelet count ≥ 100,000/μL (≥ 100 x 109/L) and haemoglobin ≥ 12 g/dL (≥ 120 g/L or ≥ 7.45 mmol/L) at the time of Screening and prior to the first dose administration.
7. Adequate hepatic function, defined as having total bilirubin ≤ 1.5x ULN (excluding Gilbert's syndrome) and AST and/or ALT ≤ 3x ULN at the time of Screening and prior to the first dose administration; no clinical signs or known laboratory OR radiographic evidence consistent with cirrhosis of the liver.
8. Adequate renal function, defined as having serum creatinine ≤ 2.5x ULN at the time of Screening and prior to the first dose administration.

Part 3 (patients who have completed Week 24 of Part 2)

1. Completed Week 24 of Part 2 with no major compliance issues.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the extension study with the Investigator or delegate.
3. Adaquate haematologic function, defined as having platelet count ≥ 100,000/μL and haemoglobin ≥ 8 g/dL (4.97 mmol/L) at Week 20 in Part 2.
4. Adequate hepatic function, defined as having total bilirubin ≤ 1.5x ULN (excluding Gilbert's syndrome) and AST and/or ALT ≤ 3x ULN at Week 20 in Part 2 with no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis.
5. Adequate renal function, defined as serum creatinine ≤ 2.5x ULN at Week 20 in Part 2.

Part 4 (Patients who have completed Week 48 of Part 3):

1. Completed Week 48 of Part 3 with no major compliance issues.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the extension study with the Investigator or delegate.
3. Adequate haematologic function, defined as platelet count ≥ 100,000/μL and haemoglobin ≥ 8 g/dL (4.97 mmol/L) at Week 44 of Part 3.
4. Adequate hepatic function, defined as total bilirubin ≤ 1.5x ULN (excluding Gilbert's syndrome) and AST and/or ALT ≤ 3 x ULN at Week 44 of Part 3 with no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis.
5. Adequate renal function, defined as serum creatinine ≤ 2.5x ULN at Week 44 of Part 3.

Part 5 (Patients who have completed Week 24 of Part 4):

1. Completed Week 24 of Part 4 with no major compliance issues.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the extension study with the Investigator or delegate.
3. Adequate haematologic function, defined as platelet count ≥ 100,000/μL and haemoglobin ≥ 8 g/dL(4.97 mmol/L) at Week 20 of Part 4.
4. Adequate hepatic function, defined as total bilirubin ≤ 1.5x ULN (excluding Gilbert's syndrome) and AST and/or ALT ≤ 3 x ULN at Week 20 of Part 4 with no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis.
5. Adequate renal function, defined as serum creatinine ≤ 2.5x ULN at Week 20 of Part 4.

Part 6 (Patients who have completed Week 52 of Part 5):

1. Completed Week 52 of Part 5 with no major compliance issues.
2. Capable of giving written informed consent to participate after reading the information and consent form, and after having the opportunity to discuss the extension study with the Investigator or delegate.
3. Adequate haematologic function, defined as platelet count ≥ 100,000/μL and haemoglobin ≥ 8 g/dL (4.97 mmol/L) at Week 48 of Part 5.
4. Adequate hepatic function, defined as total bilirubin ≤ 1.5x ULN (excluding Gilbert's syndrome) and AST and/or ALT ≤ 3 x ULN at Week 48 of Part 5 with no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis.
5. Adequate renal function, defined as serum creatinine ≤ 2.5x ULN at Week 48 of Part 5.

Exclusion Criteria:

1. Healthy subject/patient with known thrombophilia.
2. Healthy subject/patient with previous Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE), Myocardial Infarction (MI) or stroke.
3. Healthy subject/patient with uncontrolled hypertension (healthy subject: Systolic BP > 140 mmHg, Diastolic BP > 90 mmHg and patient: Systolic BP > 160 mmHg, Diastolic BP > 100 mmHg).
4. Healthy subject/patient with diagnosis of diabetes requiring drug treatment.
5. Healthy subject/patient who has active cancer or requiring therapy for cancer or diagnosis of cancer in previous 12 months before the first dose of IMP.
6. Healthy subject who has participated in a clinical trial during the 90 days prior to dosing and patient who has participated in a clinical trial during the 30 days prior to screening.
7. Healthy subject/patient with any major medical or psychological or psychiatric condition that could cause the healthy subject/patient to be unsuitable for the study or could interfere with the interpretation of the study results.
8. Healthy subject/patient with a history of or other evidence of recent alcohol or drug abuse (in the previous 12 months before the first dose of IMP).
9. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
10. Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function).
11. Donation of 450 mL or more blood within the 3 months before the first dose of IMP.

    Additional Exclusion Criteria only applicable for Part 1b, Part 2, Part 3, Part 4 and Part 5:
12. Known HIV infection with CD4 count (or T-cell count) < 200 cells/μL within 24 weeks prior to screening.
13. Any other conditions or comorbidities, which in the opinion of the investigator would make the patient unsuitable for enrolment or could interfere with participation in or completion of the study.
14. Treatment with anticoagulant or antiplatelet drugs.

Additional Exclusion Criteria only applicable for Part 3:

1. Patient is unable to tolerate SerpinPC.
2. Patient with clinically significant safety data in Part 2 as determined by the Safety Review Committee or Investigator.
3. Patient with persistent high titre antidrug antibodies (ADAs) confirmed in Part 2 (up to Week 12 or Week 16).
4. Participation in a clinical trial, except Part 2, during the 30 days prior to Day 0.

Additional Exclusion Criteria only applicable for Part 4:

1. Patient is unable to tolerate SerpinPC.
2. Patient with clinically significant safety data in Part 3 as determined by the Safety Review Committee or Investigator.
3. Participation in a clinical trial, except Part 3, during the 30 days prior to Day 0.

Additional Exclusion Criteria only applicable for Part 5:

1. Patient is unable to tolerate SerpinPC.
2. Patient with clinically significant safety data in Part 4 as determined by the Safety Review Committee or Investigator.
3. Participation in a clinical trial, except Part 4, during the 30 days prior to Day 0.

Additional Exclusion Criteria only applicable for Part 6:

1. Patient is unable to tolerate SerpinPC.
2. Patient with clinically significant safety data in Part 5 as determined by the Safety Review Committee or Investigator.
3. Participation in a clinical trial, except Part 5, during the 30 days prior to Day 0.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From Day 1 up to 74 weeks
  Number of Participants with One or More Drug Related Adverse Events (AEs) or any Serious AEs

SECONDARY OUTCOMES:
PK of SerpinPC in plasma after single dose administration - Cmax | From Day 1 up to 26 weeks
  Maximal concentration
PK of SerpinPC in plasma after single dose administration - Tmax | From Day 1 up to 26 weeks
  Time of maximal concentration
PK of SerpinPC in plasma after single dose administration - kel | From Day 1 up to 26 weeks
  Elimination rate constant
PK of SerpinPC in plasma after single dose administration - t1/2 | From Day 1 up to 26 weeks
  Terminal elimination half-life
PK of SerpinPC in plasma after single dose administration - AUC | From Day 1 up to 26 weeks
  Area under the concentration-time curve
PK of SerpinPC in plasma after single dose administration - AUC0-t | From Day 1 up to 26 weeks
  Area under the concentration-time curve from time of dosing to last measureable concentration
PK of SerpinPC in plasma after single dose administration - AUC0-inf | From Day 1 up to 26 weeks
  Area under the concentration-time curve from time of dosing extrapolated to infinity.
PK of SerpinPC in plasma after single dose administration - AUC% | From Day 1 up to 26 weeks
  Residual area under the concentration-time curve.
PK following multiple dose administration - Cmax | From Day 1 up to 26 weeks
  Maximal concentration
PK following multiple dose administration - Tmax | From Day 1 up to 26 weeks
  Time to maximal concentration
PK following multiple dose administration - Kel | From Day 1 up to 26 weeks
  Elimination rate constant
PK following multiple dose administration - t1/2 | From Day 1 up to 26 weeks
  Terminal elimination half-life
PK following multiple dose administration - AUC | From Day 1 up to 26 weeks
  Area under the concentration-time curve
PK following multiple dose administration - AUC(0-τ) | From Day 1 up to 26 weeks
  Area under the concentration-time curve from time of dosing to the end of the dosing interval
PK following multiple dose administration - R0 | From Day 1 up to 26 weeks
  Accumulation ratio
PK following multiple dose administration - Ctrough | From Day 1 up to 26 weeks
  Trough concentration

OTHER OUTCOMES:
Effect of SerpinPC on Annualised Bleeding Rate and factor usage | From Day 1 up to 26 weeks
  Descriptive statistics of actual absolute and change from baseline values will be summarized
Effect of SerpinPC on Annualised Bleeding Rate following extended monthly dosing | From Day 1 up to 74 weeks
  Descriptive statistics of actual absolute and change from baseline values will be summarized

CONTACTS AND LOCATIONS:
Locations (3):
- Arensia Clinical Research Unit, Tbilisi, Georgia
- Arensia Clinical Research Unit, Chisinau, Moldova
- Simbec Research Ltd, Merthyr Tydfil, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No